CLINICAL TRIAL: NCT03118180
Title: The Safety and Efficacy Evaluation of CD19 Targeted Chimeric Antigen Receptor T Cells for B Cell Lymphoma
Brief Title: CD19 Targeted Chimeric Antigen Receptor T Cells for B Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Innovative Cellular Therapeutics Co., Ltd. (Other)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART19-001
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART19 group (Experimental): All patients were included for CART19 therapy
  Interventions: Biological: CD19 targeted chimeric antigen receptor T cells

INTERVENTIONS:
Biological: CD19 targeted chimeric antigen receptor T cells — CD19 targeted chimeric antigen receptor T cells for refractory and relapsed B cell lymphoma

SUMMARY:
A prospective study to evaluate the safety and efficacy of CART19 for refractory/relapsed B cell lymphoma.

DETAILED DESCRIPTION:
A prospective study to evaluate the safety and efficacy of CART19 for refractory/relapsed B cell lymphoma. Complete remission rate, overall survival rate, relapse rate and CRS rate were monitored. CART associated toxicities were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed aggressive B cell lymphoma
2. Chemotherapy-refractory disease, defined as one or more of the following:

   No response to first-line therapy (primary refractory disease); PD as best response to first-line therapy SD as best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R- CHOP) with SD duration no longer than 6 months from last dose of therapy OR No response to second or greater lines of therapy PD as best response to most recent therapy regimen SD as best response after at least 2 cycles of last line of therapy with SD duration no longer than 6 months from last dose of therapy OR Refractory post-ASCT Disease progression or relapsed ≤12 months of ASCT (must have biopsy proven recurrence in relapsed subjects) if salvage therapy is given post-ASCT, the subject must have had no response to or relapsed after the last line of therapy
3. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia)
4. Age 18 or older
5. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
6. ANC ≥1000/uL
7. Platelet count ≥75,000/uL
8. Absolute lymphocyte count ≥100/uL
9. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min Serum ALT/AST ≤2.5 ULN Total bilirubin ≤1.5 mg/dl, except in subjects with Gilbert's syndrome. Cardiac ejection fraction ≥ 50% ,no evidence of pericardial effusion as determined by an ECHO, and no clinically significant ECG findings No clinically significant pleural effusion Baseline oxygen saturation >92% on room air
10. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)

Exclusion Criteria:

1. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years
2. History of Richter's transformation of CLL
3. Autologous stem cell transplant within 6 weeks of planned CAR-C19 infusion
4. History of allogeneic stem cell transplantation
5. Prior CD19 targeted therapy with the exception of subjects who received CAR-C19 in this study and are eligible for re-treatment
6. Prior chimeric antigen receptor therapy or other genetically modified T cell therapy
7. History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
8. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the K Medical Monitor.
9. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti- HCV positive). A history of treated hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
10. Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted
11. Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases
12. History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
13. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
14. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
15. Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression
16. Primary immunodeficiency
17. History of deep vein thrombosis or pulmonary embolism within 6 months of enrollment
18. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
19. History of severe immediate hypersensitivity reaction to any of the agents used in this study
20. Live vaccine ≤ 6 weeks prior to start of conditioning regimen
21. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential
22. Subjects of both genders who are not willing to practice birth control from the time of consent through 6 months after the completion of CAR-C19
23. In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
24. History of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | Up to 30 months
  the number of response patients/the number of total patients

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, Dr, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided